CLINICAL TRIAL: NCT03837860
Title: Reducing the Abuse Liability of Prescription Opioids in Recreational Drug Users: A Pilot Study
Brief Title: Reducing the Abuse of Opioids in Drug Users
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC20180167
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Opioid Abuse, Unspecified; Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxycodone; Risperidone; ziprasidone

STUDY DESIGN:
Intervention Model Description: Double-blinded, crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oxycodone/Placebo (Active Comparator): Each study participant will receive all three study interventions in random order.In this arm, the participant receives oxycodone or placebo
  Interventions: Drug: Oxycodone/Placebo
- Oxycodone/Risperidone (Active Comparator): Each study participant will receive all three study interventions in random order. In this arm the participant receives a combination of oxycodone or risperidone
  Interventions: Drug: Oxycodone/Risperidone
- Oxycodone/Ziprasidone (Active Comparator): Each study participant will receive all three study interventions in random order. In this arm the participant receives a combination of oxycodone or ziprasidone
  Interventions: Drug: Oxycodone/Ziprasidone

INTERVENTIONS:
Drug: Oxycodone/Placebo — Oxycodone 20 mg plus placebo
  Other Names: Oxycontin/Placebo
  Arms: Oxycodone/Placebo
Drug: Oxycodone/Risperidone — Oxycodone (20mg) plus Risperidone (2 mg)
  Other Names: Oxycontin/Risperdal
  Arms: Oxycodone/Risperidone
Drug: Oxycodone/Ziprasidone — Oxycodone (20mg) plus Ziprasidone (80 mg)
  Other Names: Oxycontin/Geodon
  Arms: Oxycodone/Ziprasidone

SUMMARY:
The consequences of prescription opioid abuse are serious and the number of deaths from unintended overdose have quadrupled over the last 15+ years. Opioid analgesics remain among the most commonly abused class of substances in the United States. Moreover, patients who take pain medications for legitimate reasons may develop an opioid use disorder (OUD), with as many as 1 in 4 patients becoming dependent on their pain medications. Because of changing access to prescription opioid analgesics due to an increasingly negative prescribing climate and changes in guidelines, patients often turn to heroin, with an estimated 1 in 15 pain patients trying heroin within 10 years. Pain is a symptom that can be severely debilitating and needs to be treated adequately to improve the quality of life. Clinicians, then, are in a proverbial "catch-22" situation whereby treating a patient's chronic pain also exposes them to medications with substantial abuse liability and overdose risk. In this proposal, a method aimed at reducing the abuse potential of prescription opioid medications, without altering their analgesic efficacy, is described.

The study team hypothesize that this can be accomplished by administering a fixed-dose-combination of an opioid with an atypical antipsychotic drug, in the same pill or capsule.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 21 to 65 years of age, capable of understanding and providing consent in English, and capable of complying with the outcome instruments used.
* Recreational opioid use (i.e. defined as prescription opioid use for nontherapeutic purposes on at least 10 occasions within the previous year and at least once in the 12 weeks prior to screening)
* Reported tolerated doses to opioid medications

Exclusion Criteria:

* Currently receiving pharmacotherapy for psychiatric disorder, current suicide risk, or past history of major psychiatric disorder such as bipolar disorder/psychosis
* Presence of dementia
* Current neuroleptic medication in past 30 days
* Pregnancy
* Positive drug urine test for Barbiturates, Benzodiazepines, Methadone, and Buprenorphine.
* Subjects with a prolonged QT interval greater than 430ms (i.e. QTc >430ms)
* Subjects with a heart rate of less than 60 or greater than 100bpm will be assessed by a physician for symptomatic bradycardia/tachycardia and eligibility determined on a case-by-case basis
* Subjects with serum potassium and/or magnesium outside of normal range of our institutional laboratory within the past three months from time of screening.
* Subjects who appears intoxicated on the day of study visit by an on-site physician.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Change in Bipolar Visual Analog Scale (VAS) of Drug Likability | Study visit 2 to study visit 6, an average of 10 days
  The bipolar VAS is used to measure the Change in magnitude of "drug liking". The Drug Effects Questionnaire AKA the bipolar VAS of Drug Likability is a 5 item self-administered assessment where participants place a mark on a line from 0 to 100, "strongly dislike" at 0 (on the left hand side), "no effect" at 50 (in the center) and "strongly like" at 100 (on the far right). Change from visit 2 to visit 6 will be measured.

SECONDARY OUTCOMES:
Change in Profile of Mood States (POMS) | Study visit 2 to study visit 6, an average of 10 days
  POMS is a self-administered, standard validated psychological test formulated by McNair et al. (1971). It is a used to assess transient, distinct mood states. The questionnaire contains 65 words/statements that describe feelings people have. Outcome will be assessed using categorical and continuous data analysis comparing across groups. Change from visit 2 to visit 6 will be measured.
Change in Addiction Research Center Inventory Short Form (ARCI-SF) | Study visit 2 to study visit 6, an average of 10 days
  The ARCI is a self-administered, standardized questionnaire for assessing subjective effects of psychoactive drugs that was developed in the early 1960s at the National Institute of Mental Health Addiction Research Center. For this study, we will be using the 49-item short form. Outcome will be assessed using categorical and continuous data analysis comparing across groups. Change from visit 2 to visit 6 will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ameet Nagpal, MD, Principal Investigator — UT Health San Antonio
Locations (1):
- Westgate Pain Clinic, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No